CLINICAL TRIAL: NCT01448408
Title: Evaluation of the Sensitivity, Specificity, and Test Accuracy of Corneal Biomechanical Metrics, Anterior Segment Data and a Combination Model, in Differentiating Forme Fruste Keratoconus (FFK) From Healthy Corneas.
Brief Title: Corneal Biomechanical Properties and Anterior Segment Parameters, in Forme Fruste Keratoconus
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Lecturer, Democritus University of Thrace
Other Study IDs: 26/27-09-2011
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Keratoconus; Forme Fruste Keratoconus
Keywords: Forme Fruste Keratoconus; Corneal Biomechanical properties; Anterior Segment Parameters; Diagnostic Capacity
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Forme Fruste Keratoconus group (FFKG): FFK eyes had to present a) no apparent signs of KC in clinical examination b) stage 0 in the Amsler-Krumeich scale, and c) demonstrate a KISA index value between 60-100%
- Normal Group (CG): Eligibility for participation in the CG was confirmed by consecutive topographies, while all CG participants had to present uneventful ophthalmologic history, no indications of corneal pathology in slit-lamp biomicroscopy and Placido disk-based videokeratography and KISA index value less than 60%, as well.

SUMMARY:
The present study attempts to evaluate the diagnostic capacity of a) anterior segment parameters b) biomechanical metrics and c) a combination model, in differentiating Forme Fruste Keratoconus (FFK) from healthy corneas.

The study adhered to the tenets of the Declaration of Helsinki and written informed consent was given by all participants. The study was conducted at the Eye Institute of Thrace (ΕΙΤ), in Alexandroupolis, Greece. EΙΤ is a Democritus University research institute focusing primarily on the conditions of the anterior segment of the eye.

All participants underwent a complete clinical evaluation including review of medical history, visual acuity measurements, uncorrected and best corrected visual acuity, placido disc topography, Scheimpflug camera measurements, ORA measurements , slitlamp biomicroscopy and fundoscopic examination.

All study participants were divided in two groups. The FFK group (FFKG) consisted of patients with unilateral KC.

The control group (CG) was formed by refractive surgery candidates who visited EIT's outpatients service for their preoperative examination.

CRF and CH parameters were obtained while the patient was sitting on a chair in front of the Ocular Response Analyzer (ORA; Reichert Ophthalmic Instruments, Buffalo, NY, USA) device. Upon successful fixation of the patient's eye on a red blinking target, the operator activated the device. An air puff was released by a non-contact probe, which scanned the central area of the eye and sent a signal to the ORA. In brief, the air puff causes the cornea to move inward, past applanation, and into slight concavity. After milliseconds, the air pumps shut off, the pressure decreases, and the cornea begins to return in its normal state. The system monitors the entire process and measures two pressure values, which are determined from the inward and outward applanation processes. The aforementioned measuring procedure enables the determination of CH which is related to the viscoelastic structure of the corneal tissue, and is calculated as the difference between the two pressure values at the two applanation processes, and CRF which is indicative of the overall resistance of the cornea and is calculated as a linear function of the two pressures associated with the two applanation. In order to ensure accurate results, ORA was done four times for each eye, by the same operator. Signals that differ significantly in appearance from the other signals from the same eye were deleted.

Corneal Astigmatism (Cyl), Anterior Chamber Depth (ACD), Corneal Volume at 3mm (CV3), at 5mm (CV5), and overall (CV), Central Corneal Thickness (CCT), Thinnest Corneal Thickness (TCT) and TCT co-ordinates (TCTx, TCTy) were obtained using Pentacam. KISA index was calculated using Pentacam derived topography. Pentacam is based on a rotating Scheimpflug camera and monochromatic slit light source (a blue light emitted diode at 475 nm) which rotate together. After proper alignment of the patient's head, a fixation target is shown which guides the patients gaze. A real time image of the patient's eye is shown to the examiner on the computer screen, and the image is manually focused and centered. Acceptable maps had at least 10.0mm of corneal coverage. Moreover, images with extrapolated data in the central 9.0mm zone were excluded. Regarding the measuring procedure itself, patients were asked to blink and then look at the fixation device. In case of low-quality image, the procedure was repeated until the acceptable criteria were met.

The data from the FFKG were compared with those from the CG in separate series analyses. Receiver operating characteristics (ROC) curves were applied to determine the overall predictive accuracy of the test for each studied parameter, as described by the area under the curve. We also used this approach to identify the cut-off points for studied parameters to maximize sensitivity and specificity in discriminating FFK cases from normal corneas. Logistic regression was used to support the cut-off point identified in the ROC curve analysis. We determined a cutoff value that will gave us the best predictive fit for our sample data. Furthermore, logistic regression analysis was performed to determine the predictive capability of a model that combined both corneal biomechanical properties and pentacam derived anterior segment parameters.

Differences between groups were evaluated using the Welch modified Student's two sample t-test and Mann-Whitney U test, according to normality of distribution for each parameter. A Kolmogorov-Smirnov test of normality was applied to all variables of each group. The level of significance for each parameter was set at p<0.05. The Pearson and Spearman tests were performed in order to assess correlations between anterior segment parameters and biomechanical properties, depending on their parametric evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Forme Fruste Keratoconus

Exclusion Criteria:

* previous incisional eye surgery
* corneal scars and opacities
* a history of herpetic keratitis
* severe eye dryness
* pregnancy or nursing
* current corneal infection
* underlying autoimmune disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All participants were recruited from the Outpatients Cornea service of the EIT in a consecutive if eligible basis
Sampling Method: Non-Probability Sample
Dates: Start 2007-05; Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity, Specificity and Predictive accuracy of CH, CRF, Cyl, ACD,CV, CV3, CV5 CCT, TCT, TCTx, TCTy and of a combination model
  The data from the FFKG were compared with those from the CG in separate series analysis. ROC curves were applied to determine the overall predictive accuracy of the test for each parameter. We also used this approach to identify the cut-off points for all parameters in discriminating FFK cases from normal corneas. Logistic regression was used to support the cut-off points identified in the ROC curve analysis. Furthermore, same analysis was performed to determine the predictive capability of a model that combined both corneal biomechanical properties and anterior segment parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Institute of Thrace, Alexandroupoli, Thrace, Greece